CLINICAL TRIAL: NCT03210805
Title: Investigating the Effect of 4-week Omega-3 Polyunsaturated Fatty Acid Supplementation on Inflammation
Acronym: STC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bethan Hussey (Other)
Responsible Party: Sponsor-Investigator, Bethan Hussey, Postgraduate PhD Research Student, Loughborough University
Organization: Loughborough University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R16-P138
Record Dates: First submitted 2017-07-04; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplementation (Experimental): Omega-3 Polyunsaturated Fatty Acids
  Interventions: Dietary Supplement: Omega-3 Polyunsaturated Fatty Acids Supplementation

INTERVENTIONS:
Dietary Supplement: Omega-3 Polyunsaturated Fatty Acids Supplementation — 28 days of a commercially available supplement. 4 capsules per day.
  Other Names: OmegaVia Pharmaceutical Grade Omega-3

SUMMARY:
Investigate the in vivo effects of n-3 PUFA supplementation on inflammation, gene expression and epigenetic signatures.

Ex vivo stimulation of peripheral blood mononuclear cells (PBMCs) collected pre and post n-3 supplementation and measurement of it's effect on inflammation, gene expression and epigenetic signatures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Aged between 18 and 30 years

Exclusion Criteria:

* Females (Due to differences in cell membrane incorporation of n-3 PUFAs between the sexes and the testing schedule being unable to fit in with menstrual cycle, therefore altering the blood markers that are being measured).
* Aged below 18 or above 30.
* Body mass index (BMI; in kg/ m2), below 18 or above 30.
* Use of vitamin or fish oil supplements in the last 6 months.
* High habitual oily fish consumption (<4 servings per month).
* Smoking.
* Changes in weight in the past 6 months (Dieting) or planning on changing dietary habits.
* Habitual use of anti-inflammatory drugs.
* Self-reported history of diabetes.
* History of heart disease, coagulation/bleeding disorders, metabolic disease or Serious allergy.
* Known to have blood-borne virus.
* Receipt of inoculations within 2 months of starting the study or the intention to receive such during the study.
* Donation of or intention to donate blood within 8 weeks of the first sample or at any point during the intervention.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Epigenetic regulation of Cytokine Genes | Change from Baseline at 7, 14, 21 and 28 days
  Blood Sample

SECONDARY OUTCOMES:
Total Cholesterol | Baseline, 7, 14, 21 and 28 days
  Biochemical variable
LDL (Low density lipoprotein) | Baseline, 7, 14, 21 and 28 days
  Biochemical variable
HDL (High density lipoprotein) | Baseline, 7, 14, 21 and 28 days
  Biochemical variable
Triglycerides | Baseline, 7, 14, 21 and 28 days
  Biochemical variable
Fasting Glucose | Baseline, 7, 14, 21 and 28 days
  Biochemical variable
Full Blood Count | Baseline, 7, 14, 21 and 28 days
  Biochemical variable
Height | Baseline, 7, 14, 21 and 28 days
  Standard Anthropometric Variables
Weight | Baseline, 7, 14, 21 and 28 days
  Standard Anthropometric Variables
Hip Circumference | Baseline, 7, 14, 21 and 28 days
  Standard Anthropometric Variables
Waist Circumference | Baseline, 7, 14, 21 and 28 days
  Standard Anthropometric Variables
Systolic and Diastolic Blood Pressure | Baseline, 7, 14, 21 and 28 days
  Standard Anthropometric Variables
Heart rate | Baseline, 7, 14, 21 and 28 days
  Standard Anthropometric Variables
Food Diary | Baseline, 7, 14, 21 and 28 days
  Self-reporting
Exercise Questionnaire | Baseline, 7, 14, 21 and 28 days
  Questionnaire
Ethnic background | Baseline, 7, 14, 21 and 28 days
  Questionnaire
Gene expression of Cytokine Genes | Baseline, 7, 14, 21 and 28 days
  Extracted PBMCs
ex vivo stimulation of Human Derived Blood Cells | Baseline and 28 days
  Extracted PBMCs